CLINICAL TRIAL: NCT02540460
Title: A Phase I Clinical Study, Multiple Dose of LCB01-0371 in Healthy Male Subjects
Brief Title: Multiple Ascending Dose, Phase 1 Clinical Study of LCB01-0371
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LigaChem Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: LCB01-0371-14-1-01
Record Dates: First submitted 2014-11-13; First posted 2015-09-04 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
MeSH Terms: interventions — delpazolid; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- LCB01-0371 800mg (Experimental): LCB01-0371 800mg
  Interventions: Drug: LCB01-0371 800mg; Drug: Placebo
- LCB01-0371 800mg BID (Experimental): LCB01-0371 800mg BID
  Interventions: Drug: LCB01-0371 800mg BID; Drug: Placebo
- LCB01-0371 1200mg BID (Experimental): LCB01-0371 1200mg BID
  Interventions: Drug: LCB01-0371 1200mg BID; Drug: Placebo
- Placebo (Placebo Comparator): LCB01-0371 800mg, LCB01-0371 800mg BID, LCB01-0371 1200mg BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LCB01-0371 800mg — LCB01-0371 800mg
  Arms: LCB01-0371 800mg
Drug: LCB01-0371 800mg BID — LCB01-0371 800mg BID
  Arms: LCB01-0371 800mg BID
Drug: LCB01-0371 1200mg BID — LCB01-0371 1200mg BID
  Arms: LCB01-0371 1200mg BID
Drug: Placebo — Placebo

SUMMARY:
The purpose of this study is to investigate the population pharmacokinetics of LCB01-0371 after a multiple oral dose in healthy male subjects.

To investigate safety, tolerability of LCB01-0371 after a multiple oral dose in healthy male subjects.

DETAILED DESCRIPTION:
Double blind, randomized, placebo control, multiple dose, dose escalation study

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male between 20 and 45 years of age at the time of screening
2. Subjects with body mass index (BMI) between 20 kg/m2 and 27 kg/m2 at the time of screening
3. Agree to continue to use a medically reliable dual contraception and not to donate sperm until 30th days after study completion
4. Capable of giving written informed consent, willing to participate in this clinical trial, and willing to comply with all study requirements.

Exclusion Criteria:

1. History of liver, kidney, alimentary, respiratory, musculoskeletal, endocrine, neuropsychiatric, hemato-oncologic, cardiovascular problem(s)
2. History of gastrointestinal problem (e.g. Crohn's disease, gastro-intestinal ulcer) within 6 months possibly affecting absorption of clinical trial drugs, or history of surgery (except simple appendectomy and herniotomy)
3. History of hypersensitivity reaction or history of clinically significant hypersensitivity reaction to LCB01-0371 or same class of the study drugs (linezolid) or other drugs including aspirin and antibiotics
4. History of drug abuse or positive result at urine drug screening
5. AST, ALT, r-GT, bilirubin(total) values over than 1.5 times of ULN

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
No of Adverse events | From date of randomization until follow up after 3 days from last hospital discharge

SECONDARY OUTCOMES:
Pharmacokinetics: Cmax(Peak plasma concentration) | 0(predose), 0.5, 1, 2, 4, 8 and 12hours
  Predose date: 1, 3, 6, 9, 12, 15, 17, 19, 20 and 21Days
Pharmacokinetics: AUC(Area under the curve) | 0(predose), 0.5, 1, 2, 4, 8 and 12hours
  Predose date: 1, 3, 6, 9, 12, 15, 17, 19, 20 and 21Days

CONTACTS AND LOCATIONS:
Overall Officials: Young Lag Cho, Ph.D., Study Director — Legochembioscience
Locations (1):
- Seoul National University Bundang Hospital, Bundang, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Choi Y, Lee SW, Kim A, Jang K, Nam H, Cho YL, Yu KS, Jang IJ, Chung JY. Safety, tolerability and pharmacokinetics of 21 day multiple oral administration of a new oxazolidinone antibiotic, LCB01-0371, in healthy male subjects. J Antimicrob Chemother. 2018 Jan 1;73(1):183-190. doi: 10.1093/jac/dkx367. PMID 29069400